CLINICAL TRIAL: NCT00395239
Title: The Temporal Sequence of Inflammatory Mediators During a Controlled Exacerbation of Asthma by Steroid Withdrawal.
Brief Title: Asthma/Steroid Withdrawal Study
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: This project will resume upon the completion of other research committments.
Sponsor: University of Alberta (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Irvin Mayers, Dr. Irvin Mayers, University of Alberta
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Asthma/Steroid Withdrawal
Record Dates: First submitted 2006-11-01; First posted 2006-11-02 (Estimated); Last update posted 2016-05-26 (Estimated); Status verified 2010-08

CONDITIONS: Asthma
Keywords: Asthma; Inhaled corticosteroid; ICS; Metabolites; Induced sputum; Virtual Asthma Clinic
MeSH Terms: conditions — Asthma | interventions — Fluticasone; Budesonide; ciclesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: inhaled corticosteroid

INTERVENTIONS:
Drug: inhaled corticosteroid — Fluticasone; Budesonide; Ciclesonide Dosage and frequency is patient dependant.
  Other Names: Flovent; Pulmicort; Alvesco.

SUMMARY:
The investigators propose to study the patterns of metabolite changes in subjects with asthma to determine if there is a predictable pattern prior to, and post, clinical exacerbation.

Hypothesis: 1. Metabolite profiles will change prior to detection of a clinical exacerbation in subjects with asthma.

2. There will be a measurable temporal delay before metabolite profiles return to baseline following anti-inflammatory therapy of an exacerbation of asthma.

DETAILED DESCRIPTION:
Methods:

We propose to study 20, non-smoking, asthmatic adults. Subjects will be recruited from outpatient asthma clinics in Edmonton. All subjects will meet GINA criteria for mild persistent to moderate persistent asthma. Following informed consent we will obtain blood, induced sputum and urine samples after an overnight fast and free of any caffeine for at least 24 hours. We will also obtain routine demographic information including age, sex, and usual asthma medication usage. We will obtain health related quality of life status using generic (15D) and disease specific (Asthma Quality of Life) questionnaires. Subjects will be instructed regarding use of peak flow meters and the typical symptoms associated with loss of asthma control. They will be instructed regarding accessing a dedicated asthma website that incorporates the above questions (Visit 1). There is also a place for subjects to enter twice daily peak flow measurements. The website is password protected and each subject can access only their own individualized data entry pages. A research coordinator is able to access any subject data again using a unique password. We will use this internet-based program to monitor daily PEF and daily asthma symptoms. Patients will be instructed to access the website daily and will reassessed at 2 weeks. Subjects will then be instructed to continue with their usual asthma management and to log on to the asthma website daily to record symptoms and twice daily peak flows. Only subjects meeting criteria for well controlled asthma (GOAL criteria) along with objective compliance with study protocols over 2 weeks will then be enrolled in the next phase of the study.

Phase 1. After two weeks, subjects will return (Visit 2). At this time a blood (10 ml) and urine sample will be obtained and stored for subsequent metabolomic analysis. An exhaled gas sample will be collected and analyzed for nitric oxide concentration using a sensitive chemiluminescence technique. An induced sputum sample will also be obtained using standardized protocols and cell count and differential will be determined. The remainder of the sputum sample will also be stored for subsequent analysis. All tests will be performed in the morning after an overnight fast.

Phase 2. During the second phase of the study, subjects will be instructed to reduce their controller medication (inhaled corticosteroid alone or combined inhaled corticosteroid with long acting beta 2 agonist) by 50% e.g. from 4 puffs daily to 2 puffs daily. Subjects will log on to their website daily for 4 weeks or until they experience a mild exacerbation (see definition below). If they experience a clinical exacerbation, they will be instructed to return to the hospital site where repeat blood, urine, exhaled air and sputum testing will be obtained (Visit 3a). They will be instructed to increase their controller medication and to continue with the increased steroid phase of the study. Those not experiencing a clinical exacerbation will return to the hospital site at the end of the four weeks (Visit 3b). They will have repeat blood, urine and sputum samples and will then be instructed to eliminate controller medication for four weeks or until they experience a clinical exacerbation. Those experiencing a clinical exacerbation will be treated as outlined above. Those continuing to experience clinical good control will be brought back at four weeks for repeat blood, urine, exhaled air and sputum analysis (Visit 3c). Throughout the 4-8 week period of inhaled steroid withdrawal, patients will be asked to save a urine sample three times weekly. These samples will be stored in pre-labeled containers in their freezer until picked up by the study coordinator at weekly intervals.

Phase 3. After a patient experiences a mild exacerbation or at the end of 8 weeks of steroid reduction and elimination, patients will enter the final phase of the study. At that time all patients will be instructed to increase their controller medication back to their baseline values. They will be followed for four weeks and repeat blood, urine, exhaled air and sputum samples will be obtained (Visit 4). Finally, subjects will be instructed to double their usual controller medication for four weeks after which repeat blood, urine and sputum samples will be obtained. Again, subjects will collect and store urine samples at a frequency of 3 times per week. The subjects will then be instructed to resume their usual asthma controller medication dosing and the study will be complete (Visit 5). All tests will be performed in the morning after an overnight fast.

A mild exacerbation will be defined by any one of the following events:

1. A decrease in peak flow to less than 80% of best effort for two consecutive days.
2. An increase in reliever medication (fast acting beta 2 agonist) by 50% over baseline needs for two consecutive days
3. Waking at night due to asthma on two consecutive nights A severe exacerbation will be defined as any need for additional medical contact for treatment of asthma (e.g. Emergency Room, Walk-in Clinic) or any hospital admission for asthma. The need for oral corticosteroids will also constitute a severe exacerbation. If at any point the subjects undergo a severe exacerbation, they will be examined by either their own treating physician or by one of the physicians associated with this study and appropriate escalation of treatment will be commenced. The REB will be informed of all severe exacerbations. The study coordinator and one of the study physicians will be available by pager around the clock during the course of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Non-smoker (less than 1 pack-year).
2. Age greater than 18 years old.
3. Ability to obtain informed consent.
4. Pulmonary Function Tests demonstrating greater than 12% FEV1 reversibility following beta agonist OR a methacholine challenge consistent with airways hyper-reactivity.
5. Evidence of atopy on standardized skin test battery.
6. Mild to moderate persistent asthma classification by GINA guidelines.
7. No severe exacerbations in the preceding 3 months (defined as emergency room visit, course of oral prednisone or hospitalization).
8. Access to internet.

Exclusion Criteria:

1. Unstable asthma.
2. Patient not on inhaled corticosteroids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2006-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Metabolite changes in induced sputum | 20 weeks
Metabolite changes in urine | 20 weeks

SECONDARY OUTCOMES:
Health related quality of life status | 20 weeks
Peak expiratory flow measurements | 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Irvin Mayers, MD, FRCPC, Principal Investigator — University of Alberta
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada